CLINICAL TRIAL: NCT02203253
Title: Efficacy of Thalidomide in Preventing Chemotherapy-induced Delayed Nausea and Vomiting From Highly Emetogenic Chemotherapy: a Randomized, Multicenter, Double-blind, Placebo-controlled Phase III Trial
Brief Title: Efficacy of Thalidomide in Preventing Chemotherapy-induced Delayed Nausea and Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: China Medical University, China (Other)
Collaborators: The First Hospital of Liaoning Medical University (Unknown); The First Affiliated Hospital of Dalian Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Liaoning Cancer Hospital & Institute (Other); Shengjing Hospital (Other); General Hospital of Shenyang Military Region (Other); Liaoyang Central Hospital (Other); Third People's hospital Liaoyang (Other); Petrochemical General Hospital of Liaoyang city (Unknown); Anshan Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, M.D.,PhD, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CLOG1302
Record Dates: First submitted 2014-07-23; First posted 2014-07-29 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Neoplasms
Keywords: solid tumor; chemotherapy-induced delayed nausea and vomiting; thalidomide; prevention
MeSH Terms: conditions — Neoplasms; Vomiting | interventions — Thalidomide; Palonosetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thalidomide Group (Active Comparator): Thalidomide 100 mg by mouth twice a day on days 1-5; Palonosetron 0.25 mg intravenously on day 1; Dexamethasone 12 mg by mouth or intravenously before chemotherapy on day 1 and 8 mg on days 2-4; cycle 1.
  Interventions: Drug: Thalidomide; Drug: Palonosetron and Dexamethasone
- Placebo Group (Placebo Comparator): Placebo (for Thalidomide) tablet 100 mg by mouth twice a day on days 1-5; Palonosetron 0.25 mg intravenously on day 1; Dexamethasone 12 mg by mouth or intravenously before chemotherapy on day 1 and 8 mg on days 2-4; cycle 1.
  Interventions: Drug: Placebo for thalidomide; Drug: Palonosetron and Dexamethasone

INTERVENTIONS:
Drug: Thalidomide — 100 mg by mouth twice a day on days 1-5 after chemotherapy, cycle 1
  Arms: Thalidomide Group
Drug: Placebo for thalidomide — Placebo tablet manufactured to mimic Thalidomide 25 mg tablet 100 mg by mouth twice a day on days 1-5 after chemotherapy , cycle 1
  Other Names: Placebo tablet for thalidomide
  Arms: Placebo Group
Drug: Palonosetron and Dexamethasone — Palonosetron 0.25 mg intravenously on day 1; Dexamethasone 12 mg by mouth or intravenously before chemotherapy on day 1 and 8 mg on days 2-4; cycle 1.

SUMMARY:
This study was aimed to evaluate efficacy and tolerability of thalidomide in improving prevention of chemotherapy-induced delayed nausea and vomiting in chemotherapy-naive patients after highly emetogenic chemotherapy.

DETAILED DESCRIPTION:
This is a prospective, randomized, multi-center, double-blind, placebo-controlled clinical trial, aimed to evaluate efficacy and tolerability of thalidomide in improving prevention of chemotherapy-induced delayed nausea and vomiting (CINV) in chemotherapy-naive patients after highly emetogenic chemotherapy(HEC) (cisplatin-based regimen or cyclophosphamide combination with doxorubicin/epirubicin). A total of 820 patients are planned to be enrolled into the study. Patients treating with highly emetogenic chemotherapy will be randomized into two groups, and be treated with Thalidomide+ Palonosetron+ Dexamethasone or Placebo + Palonosetron+ Dexamethasone, respectively. The primary end point is complete response rate (CRR) for delayed CINV, and the secondary end points include the safety and quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

* 18y ≤Age≤70y
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Histologically confirmed solid neoplasm
* No prior chemotherapy
* Laboratory test must meet the following criteria: hemoglobin (HGB) ≥90g/L, neutrophil count ≥1.5×109/L, platelet count ≥85×109/L, creatinine clearance rate (CCr) ≥60ml/min, total bilirubin (TBil) ≤1.5 upper normal limitation (UNL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 UNL (For patients with liver metastasis, the AST/ALT must be ≤5.0 UNL), blood glucose ≤11.1 mmol/L
* Life expectancy of at least 12 weeks
* Signed informed consent
* For women with child bearing potential, a negative serum or urine pregnancy test result should be obtained before enrollment
* Cancer patients scheduled to receive HEC regimen. The HEC regimen was defined as chemotherapy containing a 50 mg/m2 or higher dose of cisplatin, or cyclophosphamide combination with doxorubicin/epirubicin

Exclusion Criteria:

* Diabetic patients
* Pregnant or lactated women
* Patient with history of thrombosis
* Concomitant radiotherapy
* Known hypersensitivity to thalidomide, palonosetron, or dexamethasone.
* Concurrent administration of any other drug which affect antiemetic effect evaluation such as proton pump inhibitor, H2 blocker, amifostine, sedative drugs
* CHOP regiment or taxanes-based regiment
* Existing emesis within 24 hours before chemotherapy administration
* Symptomatic brain metastasis or suspected clinical brain metastasis
* Serious uncontrolled systemic illness or medical condition: congestive heart failure, unstable angina, history of documented myocardial infarction within 6 months, uncontrolled hypertension and high risk uncontrollable arrhythmias; Obvious neurological or mental abnormalities including mental disorder, epileptic dementia, which affect compliance; Uncontrolled acute infections; Uncontrolled peptic ulcer or other contraindication for corticosteroid therapy.
* Inability to take or absorb oral medicine
* Concurrent administration of any other investigational drug, or have been enrolled in other clinical trial with investigational drug treatment within the 30 days of start of study treatment
* Unsuitable for the study or other chemotherapy determined by investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
complete response rate (CRR) for delayed CINV | 120 hours

SECONDARY OUTCOMES:
Adverse Events | Up to 3 weeks
quality of life | up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, MD., PhD, Principal Investigator — China Medical University, China
Locations (11):
- China (11):
  - Anshan Tumor Hospital, Anshan, Liaoning
  - Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of Liaoning Medical University, Jinzhou, Liaoning
  - Liaoyang Central Hospital, Liaoyang, Liaoning
  - Petrochemical General Hospital of Liaoyang city, Liaoyang, Liaoning
  - Third People's hospital Liaoyang, Liaoyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - Liaoning Tumor Hospital & Institute, Shenyang, Liaoning